CLINICAL TRIAL: NCT01598038
Title: Relation Between Safety Endpoints and Everolimus Trough Blood Level in Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEVERENAL
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Renal Cell Carcinoma
Keywords: cancer; renal; Afinitor; pharmacokinetics
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afinitor (No Intervention): The recommended dose of Afinitor is 10 mg everolimus once daily, at fixed hour.Treatment should continue as long as clinical benefit is observed or until unacceptable toxicity occurs.
  In case of frail patients, treatment could be initiated at a lower daily-dose (5mg/d for example) and then increase if tolerance is acceptable.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Everolimus is determined in whole blood by validated high performance liquid chromatography with tandem mass spectrometry after protein precipitation
  Other Names: Assessment will be performed at 15 days, 1, 3 months then every three months until the end of the treatment

SUMMARY:
The investigators hypothesize everolimus toxicities are linked to pharmacokinetic variabilities of everolimus. Thus, early detection of clinical or biological risk factors will lead to personalized dosage treatment and permit a better tolerance without altering efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 year-old.
2. Histologically documented renal cell carcinoma whatever the type.
3. One or two prior therapy with cytokines and/or VEFG-ligand inhibitors are permitted.
4. Patients with an indication to receive everolimus treatment
5. Patients able and willing to give written informed consent, before the first screening procedure.

Exclusion Criteria:

1. Patients currently receiving chemotherapy or immunotherapy
2. Prior treatment with temsirolimus
3. Contraindication in everolimus :

   * Hypersensitivity to the active substance, to other rapamycin derivatives or to any of the excipients.
   * Patients with severe hepatic impairment (Child-Pugh class C)
   * Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicinal product.
4. Pregnant or breastfeeding women
5. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Find a relationship between everolimus through blood level and treatment safety. | 2 years
  We hypothesize everolimus toxicities are linked to pharmacokinetic variabilities of everolimus. Thus, early detection of clinical or biological risk factors will lead to personalised dosage treatment and permit a better tolerance without altering efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: SEVIN Emmanuel, MD, Principal Investigator — Centre François Baclesse
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Institut Gustave Roussy, Villejuif